CLINICAL TRIAL: NCT06751069
Title: Home-based Pulmonary Rehabilitation and Health Coaching in Patients With Fibrotic Interstitial Lung Disease: A Prospective Pragmatic Randomized Waitlist-Controlled Trial
Brief Title: Home-based Pulmonary Rehabilitation and Health Coaching in Patients With Fibrotic Interstitial Lung Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Teng Moua, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-007966
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Lung Fibrosis; Lung Interstitial Disease
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Randomized waitlist control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Pulmonary Rehabilitation with Health Coaching Group (Experimental): Twelve-week intervention with home-based pulmonary rehabilitation and health coaching.
  Interventions: Behavioral: Home-based Pulmonary Rehab
- Non-use Waitlist Control Observation Group (No Intervention): 12-week non-use usual care waitlist with transition to intervention group at the end of the observation period.

INTERVENTIONS:
Behavioral: Home-based Pulmonary Rehab — Participants are expected to engage in the home-based PR routine five to six days a week for the entire 12-week study period. The PR routine begins with slow upper body and timed breathing exercises, followed by two slow balance walks for 6 minutes each. The total exercise time is 24 minutes a day followed by a 4-minute mindful breathing meditation/cool down. Exercises may be modified or repeated according to baseline activity level and as conditioning improves.
  Arms: Home-based Pulmonary Rehabilitation with Health Coaching Group

SUMMARY:
The purpose of this clinical trial is to determine the impact of a home-based pulmonary rehabilitation program with health coaching on patient-reported respiratory-related quality of life and physical activity, as compared to usual care in patients with fibrotic interstitial lung disease.

DETAILED DESCRIPTION:
The fibrotic interstitial lung diseases (f-ILD) are a group of progressive and debilitating lung diseases sharing characteristics of lung scarring on imaging and restricted breathing on pulmonary function testing (PFT). Symptoms include shortness of breath, cough, and fatigue, eventually leading to deconditioning and poor quality of life. While medical therapies are available for slowing or stopping the loss of lung function, only pulmonary rehabilitation (PR) has shown a positive impact on patient-reported shortness of breath and physical activity. Unfortunately, PR may not be widely available to all patients, and some patients may become too ill to participate in traditional center-based programs.

A primary hypothesis is that modifying the content, delivery, and setting for PR in patients with f-ILD to improve access or ease of use and supporting behavior change through a health coach will have a measurable and sustained positive impact on patient well-being and quality of life as compared to no participation or non-use.

ELIGIBILITY:
IInclusion Criteria:

* F-ILD diagnosis, any disease subtype, active or prior medical treatment
* >10% fibrosis on CT imaging
* mMRC dyspnea score >1
* All racial or ethnic categories, including non-English speakers (professional translators will be engaged to support screening, enrollment, and study participation)

Exclusion Criteria:

* Inability to walk (orthopedic/neurologic/cardiac limitation causing immobility)
* Cognitive impairment or inability to understand and follow instructions
* Traditional center-based PR completed within 3 months of initial study recruitment
* Transition to hospice or end-of-life care at the time of screening
* Acute exacerbation at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
King's Brief Interstitial Lung Disease (K- BILD) | Baseline, end of intervention (3 months), and 3 months post-intervention
  Respiratory-related quality of life questionnaire
Physical activity as measured by change in mean number of steps per day | Baseline, end of intervention (3 months), and 3 months post-intervention
  Mean number of steps as measured by Actigraph monitor over 5-7 days

SECONDARY OUTCOMES:
Modified Medical Research Council (mMRC) | Baseline, end of intervention (3 months), and 3 months post-intervention
  dyspnea scale
Living with Pulmonary Fibrosis (L-PF)-Symptoms and Impacts Questionnaire | Baseline, end of intervention (3 months), and 3 months post-intervention
  Respiratory-related quality of life questionnaire
FACIT Fatigue Scale | Baseline, end of intervention (3 months), and 3 months post-intervention
  Fatigue assessment questionnaire
Leicester Cough Questionnaire (LCQ) | Baseline, end of intervention (3 months), and 3 months post-intervention
  Cough severity assessment questionnaire

OTHER OUTCOMES:
Healthcare Utilization | Six months prior to enrollment, end of intervention (3 months), and 3 months post-intervention
  Interval clinical status as reported or assessed in the medical record for clinic, urgent, emergency room visits, and hospitalizations, for all causes

CONTACTS AND LOCATIONS:
Overall Officials: Teng Moua, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No